CLINICAL TRIAL: NCT06065319
Title: Estimating Recovery in Cardiac Rehabilitation Using Mobile Health Technology and Personalized Machine Learning
Brief Title: Wearables and Cardiac Rehabilitation
Status: Active, not recruiting | Type: Observational
Sponsor: Texas A&M University (Other)
Collaborators: Ascension Health (Industry)
Responsible Party: Sponsor
Other Study IDs: R21EB028486 (NIH)
Record Dates: First submitted 2023-08-28; First posted 2023-10-03 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Cardiac Rehabilitation
Keywords: Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Comers to Cardiac Rehabilitation: Any participant that is enrolled in cardiac rehabilitation is eligible for this study.
  Interventions: Device: Wearable Sensors

INTERVENTIONS:
Device: Wearable Sensors — Participants will wear smartwatches and smartrings and this data will be used to design algorithms which seek to find associations between device data and recovery.

SUMMARY:
The goal of this study is to collect wearable sensor data that the investigators hypothesize will be useful in future algorithm development for monitoring recovering of participants enrolled in cardiac rehabilitation programs. Participants will be provided one or more smartwatches and/or smart rings to wear during a 14 week study which includes 2 weeks of baseline data collection and a 12-week, 36-session cardiac rehabilitation program. They will capture a pre-assessment 6 minute walk tests and a post-assessment 6 minute walk test. They will otherwise conduct standard cardiac rehabilitation program procedures and our sensors will capture data and sleep information throughout the study period.

DETAILED DESCRIPTION:
The goal of this study is to collect wearable sensor data that the investigators hypothesize will be useful in future algorithm development for monitoring the recovery of participants enrolled in cardiac rehabilitation programs. Participants will be provided one or more smartwatches and/or smart rings to wear during a 14 week study which includes 2 weeks of baseline data collection and a 12-week, 36-session cardiac rehabilitation program. They will capture a pre-assessment 6 minute walk tests and a post-assessment 6 minute walk test. They will otherwise conduct standard cardiac rehabilitation program procedures and our sensors will capture data and sleep information throughout the study period.

This work will use data from cardiac rehabilitation, captured from smartwatches, and data from rest/sleep, captured from smartwatches and smartrings, to see if there are trends in recovery that can be modeled. Recovery is measured as an improvement in 6 minute walk test performance over the course of cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in Cardiac Rehabilitation - eligible all-comers to Cardiac Rehabilitation
* Age 18 or older
* Native English speaker

Exclusion Criteria:

* Inability to wear one or more SmartWatches or Smartring
* Inability to walk unassisted
* Inability to participate in cardiac rehabilitation
* Inability to use a smartphone to aid in upload of remote data
* Lack of smartphone to use in the study
* There is a change in participant health such that the participant meets any of the exclusion criteria for this study during the course of the cardiac rehab sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers to cardiac rehabilitation who are capable of using smartphones for remote data collection
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in cardiac function | 12 weeks, 36 session cardiac rehabilitation
  Improvement in the 6 minute walk test performance from pre assessment to post assessment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kurian, Principal Investigator — Ascension Health
Locations (2):
- United States (2):
  - Ascension Health, Austin, Texas
  - Texas A&M University, College Station, Texas

IPD SHARING:
Plan to Share IPD: Yes
Deidentified wearable data and 6minute walk data will be made available, upon reasonable request, for other researchers
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: At the end of the study and for at least 3 years
Access Criteria: Reasonable request and data use agreement with investigators

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT06065319/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT06065319/ICF_001.pdf